CLINICAL TRIAL: NCT00943280
Title: Population Based Screening for Barrett's Esophagus in Olmsted County : A Pilot Study
Brief Title: Barrett's Esophagus in Olmsted County
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Ganapathy A. Prasad, MD, Mayo Clinic
Other Study IDs: 08-003642
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Barrett's Esophagus
Keywords: probability of patient participation in each of the Groups 1, 2 and 3.; Identification of factors predicting poor participation in screening for Barrett's esophagus.
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric, GE junction and esophagus tissue samples collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 EGD: Olmsted county residents with no history of Barrett's esophagus,who have previously completed GERQ questionnaire, randomized to EGD.
- 2 Transnasal: Olmsted county residents with no history of Barrett's esophagus,who have previously completed GERQ questionnaire, randomized to Transnasal endoscopy.
- 3 PillCam: Olmsted county residents with no history of Barrett's esophagus,who have previously completed GERQ questionnaire, randomized to PillCam.

SUMMARY:
To compare participation rates in screening for Barrett's Esophagus (BE) using sedated esophagogastroduodenoscopy (EGD), unsedated transnasal endoscopy and capsule endoscopy in a population based cohort. An age and gender stratified random sample of 300 patients from a previously defined (in terms of the presence or absence of symptoms of gastroesophageal reflux using a validated questionnaire) population based cohort from Olmsted County11, 12 using the Rochester Epidemiology Project (REP), who have not undergone endoscopy, will be randomized to undergo screening using capsule endoscopy OR transnasal endoscopy OR conventional sedated endoscopy. The investigators will compare participation rates in the three arms.

To identify factors associated with non-participation in population screening for BE. The investigators will compare demographic and clinical factors in participants and non-participants, to help predict non-participation using data from prior surveys (data has been collected on patient demographics, bowel and reflux symptoms, employment, education, somatization behavior, psychological profiles using the validated Gastroesophageal Reflux questionnaire [GERQ] and the Bowel Disease Questionnaire [BDQ]) which have been completed by all targeted subjects. This preliminary will allow us to identify barriers to screening and develop interventions to increase participation in future larger studies.

ELIGIBILITY:
Inclusion Criteria:

* Olmsted county resident

Exclusion Criteria:

* History of known BE or endoscopy within the last 5 years;
* History of progressive dysphagia;
* Known Zenker's diverticulum;
* Known epiphrenic diverticulum;
* Known or suspected intestinal obstruction;
* Cardiac pacemakers or other implanted electro-medical devices;
* Pregnancy;
* Patient expected to undergo MRI examination within 7 days after ingestion of the capsule;
* History of prior abdominal surgery of the gastrointestinal tract (other than uncomplicated appendectomy or uncomplicated cholecystectomy) within the last six months; pregnancy;
* History of recurrent epistaxis, moved from Olmsted County or deceased;
* Significant illnesses that might impair ability to complete questionnaires (e.g. metastatic cancer, major stroke); and
* Any contraindication to esophageal biopsy (such as anticoagulation using warfarin or clopidogrel [Plavix]).

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Olmsted county residents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable for this aim will be the number of subjects in each group that need to be contacted until 20 in each group agree to participate in this study. | one year

SECONDARY OUTCOMES:
To access variables for prediction of non-participation: age, gender, education level, employment, marital status, esophageal symptoms | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ganapathy A. Prasad, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Chang JY, Talley NJ, Locke GR 3rd, Katzka DA, Schleck CD, Zinsmeister AR, Dunagan KT, Wu TT, Wang KK, Prasad GA. Population screening for barrett esophagus: a prospective randomized pilot study. Mayo Clin Proc. 2011 Dec;86(12):1174-80. doi: 10.4065/mcp.2011.0396. PMID 22134936